CLINICAL TRIAL: NCT00968968
Title: A Randomized, Phase III, Open-label Study of Lapatinib Plus Trastuzumab Versus Trastuzumab as Continued HER2 Suppression Therapy After Completion of First- or Second-line Trastuzumab Plus Chemotherapy in Subjects With HER2-positive Metastatic Breast Cancer
Brief Title: Continued HER2 Suppression With Lapatinib Plus Trastuzumab Versus Trastuzumab Alone
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 112515; CLAP016A2306 (Other: Novartis)
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Cancer
Keywords: carcinoma, breast lump, Pagets disease, breast cancer positive for human epidermal growth factor receptor 2, breast cancer progression, estrogen-receptor
MeSH Terms: conditions — Neoplasms; Carcinoma | interventions — Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Lapatinib plus Trastuzumab (Experimental)
  Interventions: Drug: Lapatinib; Biological: Trastuzumab
- Arm 2: Trastuzumab (Active Comparator)
  Interventions: Biological: Trastuzumab

INTERVENTIONS:
Drug: Lapatinib — Oral Lapatinib 1000 mg once daily. Lapatinib was a small molecule, reversible inhibitor targeting HER2 tyrosine kinase receptor.
  Arms: Arm 1: Lapatinib plus Trastuzumab
Biological: Trastuzumab — IV Trastuzumab 6 mg/kg every three weeks. Trastuzumab was a humanized, monoclonal antibody directed against the extracellular domain of the HER2 tyrosine kinase receptor.

SUMMARY:
This was a randomized, open-label, multi-center Phase III study evaluating the efficacy and safety of lapatinib in combination with trastuzumab versus trastuzumab alone as continued HER2 suppression therapy in women with HER2-positive metastatic breast cancer (MBC). Eligible subjects should have completed 12 to 24 weeks of first- or second-line treatment with trastuzumab plus chemotherapy, experienced either complete disappearance of all metastatic lesions, or persistence of metastatic disease (stable disease) without unequivocal progression or the occurrence of new lesions, and been indicated to continue to receive trastuzumab alone as maintenance therapy. Eligible subjects who entered the LPT112515 study on first-line treatment should not have known history of central nervous system (CNS) metastases; subjects who entered the study on second-line treatment should not have known history of CNS metastases or have stable (asymptomatic and off steroids ≥3 months) CNS metastases. The primary objective of this study was to compare progression-free survival (PFS) in subjects with HER2-positive MBC randomized to receive treatment with lapatinib plus trastuzumab versus those randomized to receive trastuzumab alone. The secondary objectives included overall survival, clinical benefit response rate (CR, PR or SD ≥24 weeks) and the qualitative and quantitative adverse event profile of the 2 treatment arms. It was estimated that 280 subjects (140 per group) would be required to observe 193 PFS events.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form (ICF)
* Female, ≥18 years of age
* Histologically verified breast cancer with distant metastases (metastatic breast cancer)
* Documentation of HER2 overexpression or gene amplification in the invasive component of either the primary tumor or metastatic disease site defined as:
* 3+ by IHC and/or
* HER2/neu gene amplification by fluorescence, chromogenic or silver in situ hybridization [FISH, CISH or SISH; >6 HER2/neu gene copies per nucleus or a FISH, CISH or SISH HER2 gene copies to chromosome 17 signal ratio of ≥2.0]
* Completed 12 to 24 weeks of first- or second-line treatment with trastuzumab in combination with chemotherapy
* Either complete disappearance of all lesions, or persistence of metastatic disease (stable disease) without unequivocal progression or the occurrence of new lesions
* Documentation of lesion response during the course of therapy received prior to randomization (i.e., improvement or no worsening of tumor burden; the absence of new lesions)
* Measurable disease is not required for study participation
* No known or suspected (associated neurological signs and symptoms) brain metastases (including leptomeningeal involvement)
* Stable brain metastasis (defined as asymptomatic and off steroids ≥3 months) are permitted in subjects on second-line treatment (completed 12-24 weeks of second-line treatment with trastuzumab plus chemotherapy)
* Baseline of Left Ventricular Ejection Fraction (LVEF) ≥50% measured by echocardiography (ECHO) or multi-gated acquisition scan (MUGA)
* Completion of screening assessments
* Have adequate marrow and organ function

Exclusion Criteria:

* History of other malignancy. Subjects who have been disease-free for 5 years or subjects with a history of completely resected non-melanoma skin cancer (basal or squamous) are eligible
* Eastern Cooperative Oncology Group (ECOG) Performance Status >2
* Concurrent anti-cancer treatment, except anti-hormonal therapy for subjects with hormone receptor positive breast cancer
* Concurrent treatment with an investigational agent
* Prior treatment with anti-HER2 therapy, except trastuzumab or lapatinib
* Concurrent treatment with protocol-defined prohibited medications (refer to protocol for details)
* Serious cardiac illness or medical condition including but not confined to:
* Uncontrolled arrhythmias
* Uncontrolled or symptomatic angina
* History of congestive heart failure (CHF)
* Myocardial infarction <6 months from study entry
* Acute or current active (requiring anti-viral therapy) hepatic or biliary disease (with the exception of subjects with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Concurrent disease or condition that may interfere with study participation, or any serious medical disorder that would interfere with the subject's safety (for example, active or uncontrolled infection or any psychiatric condition prohibiting understanding or rendering of informed consent)
* Women of childbearing potential, including women whose last menstrual period was <12 months ago (unless surgically sterile) who are unable or unwilling to use adequate contraceptive measures during the study treatment period. Adequate contraception includes intra-uterine device, barrier methods with spermicide, or oral contraceptives (unless clinically contraindicated for the subject population or per local practice, refer to protocol for further details)
* Pregnant or lactating females
* Any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to any of the study agents or their excipients that, in the opinion of the Investigator or GSK medical monitor , contra-indicates participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-01-20 (Actual); Primary Completion 2014-02-21 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (100):
- United States (96):
  - Novartis Investigative Site, Chandler, Arizona
  - Novartis Investigative Site, Flagstaff, Arizona
  - Novartis Investigative Site, Gilbert, Arizona
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Sedona, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Pablo, California
  - Novartis Investigative Site, Santa Maria, California
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Hudson, Florida
  - Novartis Investigative Site, New Port Richey, Florida
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Dublin, Georgia
  - Novartis Investigative Site, Arlington Heights, Illinois
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Evanston, Illinois
  - Novartis Investigative Site, Glenview, Illinois
  - Novartis Investigative Site, Highland Park, Illinois
  - Novartis Investigative Site, Joliet, Illinois
  - Novartis Investigative Site, Niles, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Winfield, Illinois
  - Novartis Investigative Site, Goshen, Indiana
  - Novartis Investigative Site, Mishawaka, Indiana
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Silver Spring, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Brownstown, Michigan
  - Novartis Investigative Site, Dearborn, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, West Bloomfield, Michigan
  - Novartis Investigative Site, Burnsville, Minnesota
  - Novartis Investigative Site, Coon Rapids, Minnesota
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Fridley, Minnesota
  - Novartis Investigative Site, Maplewood, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Novartis Investigative Site, Woodbury, Minnesota
  - Novartis Investigative Site, Columbia, Missouri
  - Novartis Investigative Site, Jefferson City, Missouri
  - Novartis Investigative Site, Billings, Montana
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Cary, North Carolina
  - Novartis Investigative Site, Elizabeth City, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Washington, North Carolina
  - Novartis Investigative Site, Abington, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Radnor, Pennsylvania
  - Novartis Investigative Site, Abilene, Texas
  - Novartis Investigative Site, Beaumont, Texas
  - Novartis Investigative Site, Bedford, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Garland, Texas
  - Novartis Investigative Site, Grapevine, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Kerrville, Texas
  - Novartis Investigative Site, Odessa, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Bountiful, Utah
  - Novartis Investigative Site, Layton, Utah
  - Novartis Investigative Site, Murray, Utah
  - Novartis Investigative Site, Provo, Utah
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Sandy City, Utah
  - Novartis Investigative Site, Arlington, Virginia
  - Novartis Investigative Site, Chesapeake, Virginia
  - Novartis Investigative Site, Fairfax, Virginia
  - Novartis Investigative Site, Gainesville, Virginia
  - Novartis Investigative Site, Hampton, Virginia
  - Novartis Investigative Site, Leesburg, Virginia
  - Novartis Investigative Site, Newport News, Virginia
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Virginia Beach, Virginia
  - Novartis Investigative Site, Williamsburg, Virginia
  - Novartis Investigative Site, Edmonds, Washington
  - Novartis Investigative Site, Federal Way, Washington
  - Novartis Investigative Site, Gig Harbor, Washington
  - Novartis Investigative Site, Lakewood, Washington
  - Novartis Investigative Site, Puyallup, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Tacoma, Washington
- Canada (4):
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Rimouski, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 subjects with HER2-positive metastatic breast cancer were enrolled.
Pre-assignment Details: Subjects enrolled in the study were randomized 1:1 to either of the arms.
Groups:
- Lapatinib + Trastuzumab: Lapatinib 1000 mg oral once daily plus intravenous (iv) trastuzumab 6 mg/kg once every 3 weeks.
- Trastuzumab: Trastuzumab iv 6 mg/kg once every 3 weeks
Period: Overall Study
Arm/Group | Lapatinib + Trastuzumab | Trastuzumab
Started | 20 | 17
Completed | 4 | 3
Not Completed | 16 | 14
Not completed — Study closed/terminated | 10 | 10
Not completed — Protocol defined stopping criteria | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized subjects and based on the treatment to which the subject was randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib + Trastuzumab | Trastuzumab | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12.70) | 59.1 (9.44) | 56.5 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) with lapatinib plus trastuzumab versus trastuzumab alone.
  Progression-free survival (PFS) is defined as the time from randomization to the earliest date of disease progression (with radiological evidence) or death from any cause, or to last contact date up to 21Feb2014.
  Disease Progression was defined using Response Evaluation Criteria In Solid Tumors (RECIST v1.1), a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum diameters recorded since the treatment started (the sum must have an absolute increase from nadir of 5mm), or an unequivocal progression of existing non-target lesions, or the appearance of new lesions.
Time Frame: Time from randomization until disease progression or death, approximately 4 years
Population: Intent-to-treat population: All randomized subjects and based on the treatment to which the subject was randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib + Trastuzumab | Trastuzumab
Number analyzed (Participants) | 20 | 17
months | 25 [2.5 to 30.3] | 2 [1.9 to 6.4]

2. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the interval of time (in months) between the date of randomization and the date of death due to any cause.
Time Frame: Time from randomization until death, approximately 4 years
Population: Intent-to-treat population: All randomized subjects and based on the treatment to which the subject was randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib + Trastuzumab | Trastuzumab
Number analyzed (Participants) | 20 | 17
Months | NA [36.5 to NA] — Median and upper limit was not estimable due to few participants with events | NA [24.5 to NA] — Median and upper limit was not estimable due to few participants with events

3. Secondary Outcome: Best Overall Response
Description: The best overall response was the best response from the start of the treatment until disease progression/recurrence and was determined programmatically using investigators assessment of responses of target lesion, non-target lesion and new lesions based on RECIST v1.1. Complete Response (CR) = disappearance of all target lesion and non-target lesions if applicable, and no new lesion; Partial Response (PR) = ≥30% decrease in the sum of the longest diameter of target lesions and non-target lesion was neither complete response nor progressive disease (Non-CR/Non-PD) or not evaluable (NE); SD = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; PD = ≥ 20% increase from nadir of the target lesions or appearance of new lesion. CR and PR were confirmed responses. Confirmed CR - at least two determinations of CR at least 4 weeks apart before PD; Confirmed PR - at least two determinations of PR or better at least 4 weeks apart before PD.
Time Frame: approximately 4 years
Population: Intent-to-treat population: All randomized subjects and based on the treatment to which the subject was randomized
Measure: Number; unit: Participants
Arm/Group | Lapatinib + Trastuzumab | Trastuzumab
Number analyzed (Participants) | 20 | 17
Participants
  Complete response (CR) | 0 | 0
  Partial response (PR) | 2 | 0
  Stable disease (SD) | 1 | 2
  Non - CR/Non - PD | 4 | 3
  Progressive disease (PD) | 1 | 7
  Not evaluable (NE) | 12 | 5

4. Secondary Outcome: Clinical Benefit Response Rate (CR, PR or SD ≥24 Weeks)
Description: Clinical Benefit Rate (CBR) was defined as the percentage of patients achieving either a confirmed CR or PR at any time or maintaining SD for at least 24 weeks while on study, according to the investigator assessment of response per RECIST 1.1 criteria.
  Confirmed CR - at least two determinations of CR at least 4 weeks apart before PD; Confirmed PR - at least two determinations of PR or better at least 4 weeks apart before PD.
Time Frame: approximately 4 years
Population: Intent-to-treat population: All randomized subjects and based on the treatment to which the subject was randomized
Measure: Number (95% Confidence Interval); unit: Percentages of participants
Arm/Group | Lapatinib + Trastuzumab | Trastuzumab
Number analyzed (Participants) | 20 | 17
Percentages of participants | 10 [1.2 to 31.7] | 0 [NA to NA] — Confidence interval cannot be calculated due to insufficient number of patients with events.

5. Secondary Outcome: Adverse Event Profile of the Two Treatment Arms
Time Frame: From first dose of study treatment until 30 days after the last dose of study treatment, approximately 8 years.
Population: Safety population: All subjects who received any dose of lapatinib + trastuzumab or trastuzumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib + Trastuzumab | Trastuzumab
Number analyzed (Participants) | 18 | 16
Participants
  Any AEs | 18 | 16
  AEs related to study treatment | 16 | 7
  AEs leading to discont. of study treatment | 3 | 0
  AE leading to dose reduction | 0 | 0
  AE leading to dose interruption/delay | 11 | 2
  Any SAE | 7 | 4
  SAEs related to study treatment | 3 | 1
  Fatal SAEs | 0 | 0
  Fatal SAEs related to study treatment | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 8.5 years.
Description: From first dose of study treatment until 30 days after the last dose of study treatment
Groups:
- All Subjects: All Subjects
Arm/Group | Lapatinib + Trastuzumab | Trastuzumab | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/35
Serious Adverse Events (participants affected / at risk) | 7/18 | 4/17 | 11/35
Other Adverse Events (participants affected / at risk) | 18/18 | 16/17 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Trastuzumab (N=18) | Trastuzumab (N=17) | All Subjects (N=35)
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 2
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Trastuzumab (N=18) | Trastuzumab (N=17) | All Subjects (N=35)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0 | 1
Left atrial enlargement (Cardiac disorders) | 1 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Blepharospasm (Eye disorders) | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 1
Eye irritation (Eye disorders) | 1 | 0 | 1
Eye swelling (Eye disorders) | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0 | 1
Photopsia (Eye disorders) | 1 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 1
Vision blurred (Eye disorders) | 3 | 0 | 3
Visual impairment (Eye disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 15 | 5 | 20
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 3
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 12 | 4 | 16
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1 | 4
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 3 | 10
Asthenia (General disorders) | 2 | 0 | 2
Catheter site bruise (General disorders) | 1 | 0 | 1
Catheter site erythema (General disorders) | 1 | 0 | 1
Chills (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 8 | 1 | 9
Infusion site pain (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 2 | 1 | 3
Peripheral swelling (General disorders) | 1 | 1 | 2
Pyrexia (General disorders) | 4 | 1 | 5
Ulcer (General disorders) | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 1 | 2 | 3
Abscess limb (Infections and infestations) | 1 | 0 | 1
Breast cellulitis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 3 | 3
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 1
Ear infection (Infections and infestations) | 1 | 1 | 2
Herpes zoster (Infections and infestations) | 2 | 0 | 2
Infection (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 1
Localised infection (Infections and infestations) | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 3 | 4
Perineal abscess (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 2
Sepsis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 2 | 4
Skin infection (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 6
Urinary tract infection (Infections and infestations) | 1 | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Incision site swelling (Injury, poisoning and procedural complications) | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 3
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Immunoglobulins decreased (Investigations) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 1
Neutrophil count increased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 1 | 1 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 1
White blood cell count increased (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 6
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 3
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 4 | 0 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 2
Hypokinesia (Nervous system disorders) | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 3 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 3 | 2 | 5
Libido decreased (Psychiatric disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 2
Breast pain (Reproductive system and breast disorders) | 0 | 2 | 2
Genital rash (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 0 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 6
Rash (Skin and subcutaneous tissue disorders) | 10 | 4 | 14
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 1
Hot flush (Vascular disorders) | 3 | 1 | 4
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was closed to further enrollment since the enrollment rate would not allow the study to complete enrollment within an acceptable timeframe.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.